CLINICAL TRIAL: NCT00816881
Title: Application and Generalization of Flutter Mucus Clearance Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Zhang Xiangyu, Director, Tongji University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SHDC12007211
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; flutter; airway clearance; sputum; Physical Therapy Techniques
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): flutter mucus clearance device
  Interventions: Device: flutter mucus clearance device
- 2 (No Intervention): Observation

INTERVENTIONS:
Device: flutter mucus clearance device — five minutes every session, four sessions per day
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the clinical outcome and safety of flutter mucus clearance devices.

DETAILED DESCRIPTION:
Respiratory diseases are still increasing in elder population. Sputum detaining is a common contributing factor to acute exacerbation. The fluttering mucus clearance technique is expected to be a physical assisting therapy enhancing airway secretion clearance but need more clinical randomized control trial evidence.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary department: available to perform the device, in-hospital patients

  * Male and female
  * Age: 45 - 85 years
  * Chronic bronchitis, COPD
* Thoracic surgery department and surgical department (upper abdomen):

  * Patients with endotracheal intubation of general anesthesia
  * Age: 40-75 years

Exclusion Criteria:

* Not available to perform the procedure
* Untreated pneumothorax
* Diffusion interstitial lung disease
* Acute coronary syndrome
* Third stage hypertension
* Advanced cancer
* Severe heart, liver, renal , blood system and endocrine system dysfunction
* Noninvasive mechanical ventilation more than 6 hrs per day
* Patients with invasive ventilation and cannot weaning and extubation within 48 hours
* Active hemoptysis

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
days of fever (body temperature reach 38 degree Celsius or higher), days of antibiotics therapy, hospital length of stay, or at 28 days | one year

SECONDARY OUTCOMES:
rate of noninvasive mechanical ventilation, rate of trachea intubation, mortality due to any reason until discharge, total fees of in-hospital | one year

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xiangyu, MD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang XY, Wang Q, Zhang S, Tan W, Wang Z, Li J. The use of a modified, oscillating positive expiratory pressure device reduced fever and length of hospital stay in patients after thoracic and upper abdominal surgery: a randomised trial. J Physiother. 2015 Jan;61(1):16-20. doi: 10.1016/j.jphys.2014.11.013. Epub 2014 Dec 19. PMID 25534580